CLINICAL TRIAL: NCT01168219
Title: Phase II Study of the Addition of Azacitidine (NSC#102816) to Reduced-Intensity Conditioning Allogeneic Transplantation for Myelodysplasia (MDS) and Older Patients With AML
Brief Title: Busulfan, Fludarabine Phosphate, and Anti-Thymocyte Globulin Followed By Donor Stem Cell Transplant and Azacitidine in Treating Patients With High-Risk Myelodysplastic Syndrome and Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02053; NCI-2011-02053 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000681025; CALGB-100801; CALGB 100801 (Other: Alliance for Clinical Trials in Oncology); CALGB-100801 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia; Adult Acute Megakaryoblastic Leukemia; Adult Acute Monoblastic Leukemia; Adult Acute Monocytic Leukemia; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With Maturation; Adult Acute Myeloid Leukemia With Minimal Differentiation; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p21.3;q23.3); MLLT3-MLL; Adult Acute Myeloid Leukemia Without Maturation; Adult Acute Myelomonocytic Leukemia; Adult Erythroleukemia; Adult Pure Erythroid Leukemia; Alkylating Agent-Related Acute Myeloid Leukemia; de Novo Myelodysplastic Syndrome; Myelodysplastic Syndrome; Myelodysplastic Syndrome With Excess Blasts; Recurrent Adult Acute Myeloid Leukemia; Secondary Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts | interventions — Stem Cell Transplantation; Antilymphocyte Serum; Azacitidine; Busulfan; fludarabine phosphate; Methotrexate; merphos; Tacrolimus

ARMS (1):
- Treatment (chemotherapy and transplant) (Experimental): REDUCED-INTENSITY CONDITIONING: Patients receive fludarabine phosphate IV over 30 minutes on days -7 to -3, busulfan IV over 45 minutes on days -6 to -3, and anti-thymocyte globulin IV over 4-10 hours on days -6 to -5 (matched sibling donor [MSD]) or -6 to -4 (matched unrelated donor [MUD]).
  TRANSPLANTATION: Patients undergo allogeneic hematopoietic stem cell transplantation on day 0 or on days 0-1.
  GRAFT-VS-HOST DISEASE PROPHYLAXIS: Patients receive tacrolimus PO or IV on days -2 to 90 with taper on days 150-180. Patients also receive methotrexate IV on days 1, 3, 6 (MSD), and 11 (MUD).
  CONSOLIDATION: Beginning on day 42, patients receive azacitidine SC or IV on days 1.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Anti-Thymocyte Globulin; Drug: Azacitidine; Drug: Busulfan; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Other: Pharmacological Study; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic hematopoietic stem cell transplantation
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATS
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Other: Pharmacological Study — Correlative studies
Drug: Tacrolimus — Given PO or IV
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This phase II clinical trial is studying how well giving busulfan, fludarabine phosphate, and anti-thymocyte globulin followed by donor stem cell transplant and azacitidine works in treating patients with high-risk myelodysplastic syndrome and older patients with acute myeloid leukemia. Giving low doses of chemotherapy, such as busulfan and fludarabine phosphate, before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-vs-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving anti-thymocyte globulin before transplant and giving azacitidine, tacrolimus, and methotrexate after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if this treatment can improve 2-year progression-free survival (PFS) in patients with high risk myelodysplastic syndrome (MDS) and in patients with acute myeloid leukemia (AML) >= 60 yrs age

SECONDARY OBJECTIVES:

I. To determine the safety and feasibility of using post-transplantation azacitidine.

II. To determine the ability to use pharmacokinetic-directed busulfan to achieve area under the curve (AUC) within 20% of target AUC in > 80% of patients.

III. To determine the rate of grade II-IV and III-IV acute graft-vs-host disease (GVHD).

IV. To determine the incidence of extensive chronic GVHD. V. To determine treatment-related mortality at 100 days and at 1 year. VI. To determine 5-year overall survival.

OUTLINE:

REDUCED-INTENSITY CONDITIONING: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -7 to -3, busulfan IV over 45 minutes on days -6 to -3, and anti-thymocyte globulin IV over 4-10 hours on days -6 to -5 (matched sibling donor [MSD]) or -6 to -4 (matched unrelated donor [MUD]).

TRANSPLANTATION: Patients undergo allogeneic hematopoietic stem cell transplantation on day 0 or on days 0-1.

GRAFT-VS-HOST DISEASE PROPHYLAXIS: Patients receive tacrolimus orally (PO) or IV on days -2 to 90 with taper on days 150-180. Patients also receive methotrexate IV on days 1, 3, 6 (MSD), and 11 (MUD).

CONSOLIDATION: Beginning on day 42, patients receive azacitidine subcutaneously (SC) or IV on days 1-5.

Treatment repeats every 4 weeks for 6 courses. Blood and bone marrow samples may be collected periodically for correlative and pharmacokinetic studies.

After completion of study treatment, patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Meets one of the following sets of criteria:

  * Myelodysplastic syndromes (MDS):

    * Disease with high-risk features (found either at diagnosis or before initiation of cytotoxic therapy), defined as one of the following:

      * International prognostic scoring system (IPSS) risk >= intermediate-2
      * Refractory anemia with excess blasts by French-American-British (FAB) classification
      * High-risk cytogenetics (either complex or -7)
    * Less than 10% bone marrow blasts as determined by bone marrow biopsy within the past 4 weeks (reduction in marrow blast percentage may be achieved with chemotherapy or other therapy)
    * Less than 75 years old
  * Acute myeloid leukemia (AML):

    * No FAB M3
    * No acute leukemia following blast transformation of prior chronic myelogenous leukemia or other myeloproliferative disease
    * Patients with preceding MDS or treatment-related AML are eligible
    * Prior central nervous system (CNS) involvement is allowed provided the disease is in remission at transplantation
    * Morphologic complete remission (leukemia-free state) is defined as meeting all of the following criteria:

      * Bone marrow blasts < 5% (as determined by bone marrow within the past 4 weeks), but without requirement for normal peripheral blood counts
      * No extramedullary leukemia
      * No blasts in peripheral blood
    * Achieved complete remission (CR) after no more than 2 courses of induction chemotherapy

      * Patients treated with azacitidine or decitabine who achieve a leukemia-free state are eligible (may have required up to 4 courses of therapy to reach this status)
    * Age 60 to 74 years
* Donors must meet the following criteria:

  * One of the following:

    * HLA-identical sibling (6/6) by serologic typing for class (A, B) and low-resolution molecular typing for class II (DRB1)
    * Matched unrelated donor (8/8) by high-resolution molecular typing at HLA-A, -B, -C, and DRB1
  * No syngeneic donors
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Calculated creatinine clearance ≥ 40 mL/min
* Bilirubin < 2 mg/dL OR bilirubin 2-3 mg/dL provided direct bilirubin is normal
* Aspartate aminotransferase (AST) < 3 times upper limit of normal
* Diffusing capacity of the lung for carbon monoxide (DLCO) > 40% with no symptomatic pulmonary disease
* Left ventricle ejection fraction (LVEF) >= 30% by echocardiogram (ECHO) or multigated acquisition (MUGA)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled diabetes mellitus or active serious infections
* No known hypersensitivity to E. coli-derived products, azacitidine, or mannitol
* No human immunodeficiency virus (HIV) infection or active hepatitis B or C
* Prior azacitidine or decitabine allowed

  * No patients who progressed from MDS to AML during treatment with azacitidine or decitabine
* At least 4 weeks since prior deoxyribonucleic acid (DNA)-hypomethylating chemotherapy, radiotherapy, and/or surgery
* No more than 2 courses of consolidation therapy before transplantation (for patients with AML)

  * Any consolidation regimen that does not require transplantation can be used
  * No more than 6 months from documentation of morphologic CR to transplantation

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-07-15 (Actual); Primary Completion 2015-11-14 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (17):
- United States (17):
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - AdventHealth Orlando, Orlando, Florida
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Derived] Vij R, Le-Rademacher J, Laumann K, Hars V, Owzar K, Shore T, Vasu S, Cashen A, Isola L, Shea T, DeMagalhaes-Silverman M, Hurd D, Meehan K, Beardell F, Devine S. A Phase II Multicenter Study of the Addition of Azacitidine to Reduced-Intensity Conditioning Allogeneic Transplant for High-Risk Myelodysplasia (and Older Patients with Acute Myeloid Leukemia): Results of CALGB 100801 (Alliance). Biol Blood Marrow Transplant. 2019 Oct;25(10):1984-1992. doi: 10.1016/j.bbmt.2019.06.007. Epub 2019 Jun 15. PMID 31212080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2010 and October 2013, a total of 68 participants were recruited to this study.
Period: Overall Study
Arm/Group | Treatment (Chemotherapy and Transplant)
Started | 68
Completed | 63
Not Completed | 5
Not completed — off study before starting treatment | 2
Not completed — withdrew before transplant | 1
Not completed — ineligible due to CML | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy and Transplant)
Number analyzed (Participants) | 68
Age, Continuous [Median (Full Range); unit: years] | 62.9 [44.8 to 74.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 60
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68
Disease type [Count of Participants; unit: Participants]
  Myelodysplastic Syndrome (MDS) | 24
  Acute Myeloid Leukemia (AML) | 44

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival rate (percentage) at 2 and 5 years is defined as the percentage of patients who are alive and progression free at 2 and 5 years from date of transplantation respectively.
  AML progression is defined as:
  * Reappearance of leukemia blast cells in peripheral blood and > 5% blasts in marrow
  * If no circulating blasts, but the marrow contains 5-20% blasts, a repeat bone marrow >= 1 week later with > 5% blasts
  * Development of extramedullary leukemia MDS progression is defined as
  * For patients with <5% bone marrow blasts: ≥50% increase in blasts to >5% blasts
  * For patients with 5-10% bone marrow blasts: ≥50% increase to >10% blasts
  * Any of the following: Reappearance of prior documented characteristic cytogenetic abnormality or refractory cytopenias with unequivocal evidence of dysplasia on bone marrow biopsy/aspirate
Time Frame: Up to 5 years
Population: Patients who received transplant were evaluable for the primary endpoint.
Measure: Number (80% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Chemotherapy and Transplant)
Number analyzed (Participants) | 63
percentage of patients
  PFS at 2 years | 41.2 [33.9 to 49.9]
  PFS at 5 years | 26.9 [20.4 to 35.5]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival rate (percentage) at 2 and 5 years is defined as the percentage of patients who are still alive 2 and 5 years after date of transplantation respectively. Estimated using the Kaplan-Meier product limit estimator.
Time Frame: Up to 5 years
Population: Patients who received transplant were evaluable for this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Chemotherapy and Transplant)
Number analyzed (Participants) | 63
percentage of patients
  OS at 2 years | 45.7 [34.9 to 59.9]
  OS at 5 years | 31.2 [21.3 to 45.8]

3. Secondary Outcome: 100-day Mortality
Description: The number of death reported within the first 100 days after transplant.
Time Frame: Up to 100 days post-treatment
Population: Patients who received transplant and died are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Transplant)
Number analyzed (Participants) | 63
Participants | 10

ADVERSE EVENTS:
Description: 2 patients who cancelled prior to receiving any study treatment are excluded from this analysis
Arm/Group | Treatment (Chemotherapy and Transplant)
All-Cause Mortality (participants affected / at risk) | 42/66
Serious Adverse Events (participants affected / at risk) | 22/66
Other Adverse Events (participants affected / at risk) | 61/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy and Transplant) (N=66)
Anemia (Blood and lymphatic system disorders) | 18 (19)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Cardiac arrest (Cardiac disorders) | 2 (2)
Conduction disorder (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 7 (7)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1)
Growth accelerated (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 4 (4)
Scleral disorder (Eye disorders) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 12 (13)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 6 (7)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 11 (13)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (9)
Chills (General disorders) | 4 (4)
Death NOS (General disorders) | 1 (1)
Edema face (General disorders) | 2 (2)
Edema limbs (General disorders) | 10 (12)
Edema trunk (General disorders) | 3 (3)
Fatigue (General disorders) | 12 (13)
Fever (General disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2)
Hypothermia (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (2)
Pain (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 6 (6)
Lung infection (Infections and infestations) | 6 (7)
Mucosal infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 5 (5)
Alanine aminotransferase increased (Investigations) | 11 (11)
Alkaline phosphatase increased (Investigations) | 10 (10)
Aspartate aminotransferase increased (Investigations) | 11 (11)
Blood bilirubin increased (Investigations) | 7 (7)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 10 (11)
Ejection fraction decreased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Fibrinogen decreased (Investigations) | 2 (2)
INR increased (Investigations) | 3 (3)
Investigations - Other, specify (Investigations) | 3 (9)
Lymphocyte count decreased (Investigations) | 5 (5)
Neutrophil count decreased (Investigations) | 10 (11)
Platelet count decreased (Investigations) | 16 (17)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 5 (7)
White blood cell decreased (Investigations) | 8 (8)
Acidosis (Metabolism and nutrition disorders) | 3 (4)
Alkalosis (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (15)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 11 (12)
Hyponatremia (Metabolism and nutrition disorders) | 9 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (6)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 6 (6)
Encephalopathy (Nervous system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypersomnia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4)
Confusion (Psychiatric disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (9)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 9 (9)
Hypotension (Vascular disorders) | 10 (12)
Thromboembolic event (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy and Transplant) (N=66)
Anemia (Blood and lymphatic system disorders) | 58 (219)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 21 (24)
Hemolysis (Blood and lymphatic system disorders) | 1 (5)
Leukocytosis (Blood and lymphatic system disorders) | 4 (5)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 8 (21)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 15 (20)
Sinus tachycardia (Cardiac disorders) | 17 (28)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Hearing impaired (Ear and labyrinth disorders) | 3 (13)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (2)
Endocrine disorders - Other, specify (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 1 (7)
Blurred vision (Eye disorders) | 18 (45)
Cataract (Eye disorders) | 2 (4)
Conjunctivitis (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 10 (21)
Eye disorders - Other, specify (Eye disorders) | 8 (8)
Eye pain (Eye disorders) | 4 (5)
Glaucoma (Eye disorders) | 2 (9)
Photophobia (Eye disorders) | 2 (2)
Scleral disorder (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (4)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 5 (6)
Abdominal distension (Gastrointestinal disorders) | 5 (8)
Abdominal pain (Gastrointestinal disorders) | 23 (36)
Anal pain (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (6)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 32 (54)
Diarrhea (Gastrointestinal disorders) | 52 (87)
Dry mouth (Gastrointestinal disorders) | 19 (42)
Dyspepsia (Gastrointestinal disorders) | 11 (28)
Dysphagia (Gastrointestinal disorders) | 10 (10)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 9 (15)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 12 (22)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 4 (4)
Hemorrhoids (Gastrointestinal disorders) | 6 (7)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 47 (56)
Nausea (Gastrointestinal disorders) | 48 (111)
Oral hemorrhage (Gastrointestinal disorders) | 7 (7)
Oral pain (Gastrointestinal disorders) | 11 (14)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 3 (4)
Rectal ulcer (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 40 (57)
Chills (General disorders) | 21 (30)
Edema face (General disorders) | 7 (8)
Edema limbs (General disorders) | 24 (56)
Edema trunk (General disorders) | 3 (3)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 50 (155)
Fever (General disorders) | 26 (28)
Flu like symptoms (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 5 (5)
Infusion related reaction (General disorders) | 5 (7)
Injection site reaction (General disorders) | 8 (13)
Localized edema (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Neck edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 12 (16)
Pain (General disorders) | 11 (20)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 3 (10)
Immune system disorders - Other, specify (Immune system disorders) | 1 (4)
Bladder infection (Infections and infestations) | 3 (4)
Bronchial infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 29 (46)
Lip infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 6 (8)
Meningitis (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 6 (16)
Nail infection (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 3 (3)
Rash pustular (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 5 (7)
Sinusitis (Infections and infestations) | 1 (4)
Skin infection (Infections and infestations) | 3 (3)
Soft tissue infection (Infections and infestations) | 2 (3)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 7 (8)
Urinary tract infection (Infections and infestations) | 4 (5)
Bruising (Injury, poisoning and procedural complications) | 12 (21)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 7 (15)
Alanine aminotransferase increased (Investigations) | 40 (99)
Alkaline phosphatase increased (Investigations) | 23 (48)
Aspartate aminotransferase increased (Investigations) | 36 (90)
Blood bilirubin increased (Investigations) | 21 (26)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 35 (74)
Fibrinogen decreased (Investigations) | 1 (1)
GGT increased (Investigations) | 3 (10)
INR increased (Investigations) | 6 (11)
Investigations - Other, specify (Investigations) | 4 (32)
Lymphocyte count decreased (Investigations) | 28 (92)
Neutrophil count decreased (Investigations) | 56 (115)
Platelet count decreased (Investigations) | 56 (194)
Weight gain (Investigations) | 3 (5)
Weight loss (Investigations) | 20 (44)
White blood cell decreased (Investigations) | 35 (77)
Anorexia (Metabolism and nutrition disorders) | 39 (91)
Dehydration (Metabolism and nutrition disorders) | 8 (9)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 54 (156)
Hyperkalemia (Metabolism and nutrition disorders) | 24 (36)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 5 (5)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 38 (69)
Hypocalcemia (Metabolism and nutrition disorders) | 40 (64)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (6)
Hypokalemia (Metabolism and nutrition disorders) | 33 (45)
Hypomagnesemia (Metabolism and nutrition disorders) | 41 (104)
Hyponatremia (Metabolism and nutrition disorders) | 36 (72)
Hypophosphatemia (Metabolism and nutrition disorders) | 18 (22)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 12 (37)
Obesity (Metabolism and nutrition disorders) | 1 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (21)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (29)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (10)
Buttock pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 21 (41)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 11 (22)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (12)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (31)
Akathisia (Nervous system disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (3)
Dizziness (Nervous system disorders) | 16 (24)
Dysgeusia (Nervous system disorders) | 25 (51)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 29 (42)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 4 (4)
Memory impairment (Nervous system disorders) | 2 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 5 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 13 (36)
Presyncope (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 3 (4)
Somnolence (Nervous system disorders) | 3 (3)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Transient ischemic attacks (Nervous system disorders) | 1 (2)
Tremor (Nervous system disorders) | 13 (20)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (3)
Anxiety (Psychiatric disorders) | 18 (39)
Confusion (Psychiatric disorders) | 13 (14)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 11 (35)
Hallucinations (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 24 (54)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 12 (23)
Bladder spasm (Renal and urinary disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (3)
Cystitis noninfective (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 6 (6)
Proteinuria (Renal and urinary disorders) | 3 (4)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3 (4)
Renal calculi (Renal and urinary disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 10 (18)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 5 (6)
Urinary tract obstruction (Renal and urinary disorders) | 1 (2)
Urinary tract pain (Renal and urinary disorders) | 7 (8)
Urinary urgency (Renal and urinary disorders) | 4 (4)
Genital edema (Reproductive system and breast disorders) | 3 (3)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 3 (3)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (2)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 (11)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (30)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 29 (52)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 (21)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 16 (24)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (16)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (43)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5 (11)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Nail loss (Skin and subcutaneous tissue disorders) | 3 (9)
Pain of skin (Skin and subcutaneous tissue disorders) | 6 (8)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 31 (50)
Purpura (Skin and subcutaneous tissue disorders) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 34 (58)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 20 (55)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 (25)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (10)
Skin ulceration (Skin and subcutaneous tissue disorders) | 8 (12)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 40 (106)
Hypotension (Vascular disorders) | 21 (39)
Phlebitis (Vascular disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 7 (21)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less